CLINICAL TRIAL: NCT05105607
Title: A Phase 1 Open-Label Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of D-4517.2 (Hydroxyl Dendrimer VEGFR Tyrosine Kinase Inhibitor) After Subcutaneous Administration in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of D-4517.2 After Subcutaneous Administration in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ashvattha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-4517-001
Record Dates: First submitted 2021-10-26; First posted 2021-11-03 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema
Keywords: D-4517.2; Neovascular Age-related Macular Degeneration; Diabetic Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1: 0.25 mg/kg D-4517.2 (Experimental): Participants will be administered a single dose of 0.25 mg/kg D-4517.2. A sentinel participant will be enrolled for each cohort. After the sentinel participant completes Day 3, the safety review committee (SRC) will determine if it is safe to continue with the enrollment of the remaining 3 participants in the cohort. The SRC will also determine the dose escalation to the next cohort.
  Interventions: Drug: D-4517.2
- Cohort 2: 0.5 mg/kg D-4517.2 (Experimental): Participants will be administered a single dose of 0.5 mg/kg D-4517.2. A sentinel participant will be enrolled for each cohort. After the sentinel participant completes Day 3, the SRC will determine if it is safe to continue with the enrollment of the remaining 3 participants in the cohort. The SRC will also determine the dose escalation to the next cohort.
  Interventions: Drug: D-4517.2
- Cohort 3: 1.0 mg/kg D-4517.2 (Experimental): Participants will be administered a single dose of 1.0 mg/kg D-4517.2. A sentinel participant will be enrolled for each cohort. After the sentinel participant completes Day 3, the SRC will determine if it is safe to continue with the enrollment of the remaining 3 participants in the cohort. The SRC will also determine the dose escalation to the next cohort.
  Interventions: Drug: D-4517.2
- Cohort 4: 2.0 mg/kg D-4517.2 (Experimental): Participants will be administered a single dose of 2.0 mg/kg D-4517.2. A sentinel participant will be enrolled for each cohort. After the sentinel participant completes Day 3, the SRC will determine if it is safe to continue with the enrollment of the remaining 3 participants in the cohort.
  Interventions: Drug: D-4517.2

INTERVENTIONS:
Drug: D-4517.2 — Subcutaneous (SC) injection

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of D-4517.2 after single subcutaneous (SC) doses in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy man or woman age 18 to 65 years, inclusive, at the Screening Visit;
2. Has the ability to understand and sign the written informed consent form (ICF) and local medical privacy authorization forms, which must be obtained prior to any study related procedures being completed;
3. Body mass index (BMI) between 18 and 32 kg/m^2, inclusive, with body weight ≤ 100 kg;
4. Is in general good health, based upon the results of a medical history assessment, physical examination, vital signs, and laboratory profile, as judged by the Investigator;
5. Female participants of non-childbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before the Screening Visit) or postmenopausal, defined as spontaneous amenorrhea for at least 1 years, with follicle-stimulating hormone (FSH) in the postmenopausal range at screening, based on the central laboratory's ranges;
6. Female participants of childbearing potential (i.e., ovulating, premenopausal, and not surgically sterile) and all male participants must use a medically accepted contraceptive regimen (including hormonal contraceptives) during their participation in the study and for 30 days after the last administration of study drug. Medically accepted contraceptive methods are defined as those with 90% or greater efficacy;
7. Acceptable methods of contraception for male participants enrolled in the study include the following:

   • Condoms or surgical sterilization of participant at least 26 weeks before the Screening Visit (vasectomy);

   Acceptable methods of contraception for female participants enrolled in the study include the following:
   * Surgical sterilization of participant at least 26 weeks before the Screening Visit (includes hysterectomy or bilateral tubal ligation, oophorectomy, or salpingectomy);
   * Intrauterine device for at least 4 weeks before the Screening Visit; or
   * Hormonal contraception (oral, implant, injection, ring, or patch) for at least 4 weeks before the Screening Visit;
8. If male, participants must agree to abstain from sperm donation through 90 days after administration of the last dose of study drug;
9. Female participants may not be pregnant, lactating, or breastfeeding;
10. Female participants of childbearing potential must have negative result for pregnancy test at screening and Check-in;
11. Participants must have a negative test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVab), and human immunodeficiency virus (HIV) antibody at screening;
12. Participants must have an estimated glomerular filtration rate (eGFR) of ≥60 mL/min/1.73m^2 at screening;
13. Participants must have a negative urine test for drugs of abuse, cotinine, and breath alcohol test at screening and Check-in; and
14. Participants must be willing and able to abide by all study requirements and restrictions.

Exclusion Criteria:

1. Evidence of clinically significant hematologic, renal, endocrine, pulmonary, cardiac, gastrointestinal (GI), hepatic, psychiatric, neurologic, immunologic, allergic disease (including multiple or clinically significant drug allergies), or any other condition that, in the opinion of the Investigator, might significantly interfere with the absorption, distribution, metabolism, or excretion of study drug, or place the participant at an unacceptable risk as a participant in this study;
2. Evidence of systemic inflammation as measured by C-reactive protein above the upper limit of normal as measured by local lab;
3. History of malignancy (other than successfully treated basal cell or squamous cell skin cancer);
4. History or presence of an abnormal ECG that, in the opinion of the Investigator, is clinically significant;
5. Laboratory results (serum chemistry, hematology, coagulation, and urinalysis) outside the normal range at screening and Check-in and considered clinically significant in the opinion of the Investigator. Any elevation of aspartate transaminase (AST) and alanine transaminase (ALT) above the upper limit of normal at screening and/or Check-in is exclusionary. One retest of an exclusionary laboratory result is allowed at the discretion of the Investigator;
6. Has had an acute illness considered clinically significant by the Investigator within 30 days prior to screening;
7. History of alcoholism or drug abuse within 2 years prior to screening;
8. Has used any product containing nicotine within 90 days prior to screening or intends to use any product containing nicotine during the course of the study;
9. Has had any immunizations (live vaccines) in the 4 weeks prior to screening; COVID-19 vaccination within 7 days of Day 1;
10. Has used medications that affect GI motility or gastric emptying; such as metoclopramide, proton pump inhibitors, and H2 blockers; within 30 days prior to Day 1;
11. Has used any prescription or over-the-counter medication (with exception of acetaminophen), vitamins/herbal supplements (with the exception of hormonal contraceptives) within 14 days prior to Day 1;
12. Has used any other study drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to Day 1;
13. Has lost or donated >450 mL of whole blood or blood products within 30 days prior to screening;
14. Investigator has reason to believe that the participant may be unable to fulfill the protocol visit schedule or requirements;
15. Has any finding that, in the view of the Investigator or Medical Monitor, would compromise the participant's safety requirements; or
16. Is employed by the Sponsor, the Contract Research Organization (CRO), or the study site (permanent, temporary contract worker, or designee responsible for the conduct of the study), or is a family member (spouse, parent, sibling, or child) of the Sponsor, CRO, or study site employee.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Day 1 up to Day 15

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of D-4517.2 | Day 1 up to Day 3
Time to Maximum Plasma Concentration (tmax) of D-4517.2 | Day 1 up to Day 3
Apparent Terminal Rate Constant (kel) of D-4517.2 | Day 1 up to Day 3
Apparent Elimination Half-life (t1/2) of D-4517.2 | Day 1 up to Day 3
Area Under the Concentration-time Curve Based On the Last Measurable Concentration (AUC0-t) | Day 1 up to Day 3
Area Under the Concentration-time Curve from Time Zero to Infinity (AUC0-inf) | Day 1 up to Day 3
Clearance (CL) of D-4517.2 | Day 1 up to Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network (Brisbane), Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No